CLINICAL TRIAL: NCT05571527
Title: Comparison of Vaginal Hyaluronic Acid Treatment Over Autologous Platelet Rich Plasma Treatment for Genitourinary Syndrome of Menopause
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ozan Karadeniz, Principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KanuniSSEAH3
Record Dates: First submitted 2022-10-04; First posted 2022-10-07 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Genitourinary Syndrome of Menopause
Keywords: genitourinary syndrome; menopause; platelet rich plasma; vaginal atrophy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Menopause patients having genitourinary syndrome (PRP) (Experimental): Preparation of PRP sample from the patient's own blood and then the volume immediately above the erythrocyte layer was collected. Calcium gluconate in conc. 1:9 will be used as an activator. After activation, in a period of less than 2 min, approximately 4 ml of the PRP will be injected into the vaginal wall. ( at 3,6 and 9 o clock)It will be repeated once a month for 3 times.
  Interventions: Biological: Platelet Rich Plasma treatment
- vaginal hyluronic acid supplement for GSM (Active Comparator): Patients receive Vaginal Hyaluronic Acid supplement for 10 days, then once a week for 3 months.
  Interventions: Drug: Vaginal Hyaluronic Acid supplement

INTERVENTIONS:
Biological: Platelet Rich Plasma treatment — Patients receive platelet-rich plasma via injection into the vaginal area.
  Arms: Menopause patients having genitourinary syndrome (PRP)
Drug: Vaginal Hyaluronic Acid supplement — Patients receive Vaginal Hyaluronic Acid supplement for 10 days, then once a week for 3 months.
  Arms: vaginal hyluronic acid supplement for GSM

SUMMARY:
Genitourinary syndrome of menopause (GSM) is a collection of symptoms and signs caused by hypoestrogenic changes to the labia majora/minora, clitoris, vestibule/introitus, vagina, urethra, and bladder that occur in menopausal patients.

Platelet-rich plasma is produced by collecting approximately 60-90 ml (4-6 tablespoons) of blood from the vein in patient's arm. The blood is spun using a centrifuge that separates the plasma and red blood cells.

The treatment included vaginal estrogen supplement, vaginal hyaluronic acid supplement, vaginal laser, platelet-rich plasma, etc. The observational cohort study will be used for the study design. Questionnaires, pelvic examination, vaginal pap smear with maturation index (MI), vaginal pH, and other methods will be used to evaluate the effectiveness and side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

To determine the safety and feasibility of using platelet-rich plasma (PRP) treatment in menopausal patients with genitourinary syndrome

SECONDARY OBJECTIVE:

To determine the preliminary efficacy in the treatment of vaginal atrophy, urinary symptoms, assessment of sexual function, quality of life symptoms

VSQ, Vaginal health index, Vaginal maturation index, and Day-to-Day Impact of Vaginal Aging score will be used for assessments.

OUTLINE:

Patients receive platelet-rich plasma via injection into the vaginal area after obtaining plasma into PRP tubes

After 3 sessions of PRP treatment, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Women with menopause
* Patients with symptoms of genitourinary syndrome of menopause

Exclusion Criteria:

* Genitourinary bleeding or infection without a definitive diagnosis
* Coagulopathy
* Allergy to medication or therapy related to the treatment
* Chronic disease that might influence the outcome
* Using medication that might influence the outcome in 30 days
* Using hormone or steroid within 8 weeks
* Personal history of vulvovaginal conditions such as lichen sclerosis, lichen planus, vulvovaginal condyloma, vaginal intraepithelial neoplasia, vaginal carcinoma, history of cervical or other gynecologic cancer, radical pelvic surgery, acute or recurrent urinary tract infection, genital infection, history of vaginal or pelvic radiation
* Chronic pelvic pain, current pelvic tension myalgia/muscle hypertonicity
* Pelvic organ prolapse greater than stage II
* Pelvic surgery within 6 months
* Known allergy to lidocaine or prilocaine
* Use of vaginal moisturizers, lubricants, or homeopathic preparations within 2 weeks of therapy
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal health index score (VHIS) | [ Time Frame: 6 months after intervention ]
  evaluation of vaginal elasticity, secretions, pH, the presence of petechiae on the epithelial mucosa, and hydration
The Vulvovaginal Symptom Questionnaire (VSQ) | [ Time Frame: 6 months after intervention ]
  symptoms, emotions, life-impact, and sexual impact of vulvovaginal symptoms.
Day-to-Day Impact of Vaginal Aging Questionnaire | [ Time Frame: 6 months after intervention ]
  Measure of the Impact of Vaginal Symptoms on Functioning and Well-being in Postmenopausal Women
vaginal maturation index | [ Time Frame: 6 months after intervention ]
  objective, qualitative assessment of vaginal response to hormones as well as overall hormonal environment.
vaginal health index | [ Time Frame: 6 months after intervention ]
  clinical tool that, by evaluating 5 parameters (vaginal elasticity, vaginal secretions, pH, epithelial mucous membrane, vaginal hydration)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)